CLINICAL TRIAL: NCT03876834
Title: Influence of Respiratory Training on Functional Capacity in Patients With Leukemia
Brief Title: Respiratory Training in Patients With Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201617032.4
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Leukemia
Keywords: leukemia; chemotherapy; respiratory training
MeSH Terms: conditions — Leukemia | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (group A) (Experimental): Group (A) included 30 leukemic patients receiving chemotherapy in addition to training by inspiratory muscle trainer(IMT) for 4 weeks, 5 sessions /week
  Interventions: Other: respiratory training
- control group (B) (No Intervention): Group (B) included 10 leukemic patients receiving chemotherapy only

INTERVENTIONS:
Other: respiratory training — Respiratory training was done by using threshold inspiratory muscle trainer(Respironics, New Jersey , USA, No.8373-0730)
  Arms: study group (group A)

SUMMARY:
Forty male leukemic patients receiving chemotherapy were selected from National Cancer Institute, They were randomly assigned into two groups. Group (A) included 30 patients who were trained by Inspiratory muscle trainer for 4 weeks ;5 sessions/week and Group (B) included 10 patients as a control group.

The following measures were taken before and after the study period : Maximum voluntary ventilation(MVV) , 2 min walk test, FACT-G questionnaire

DETAILED DESCRIPTION:
Forty male leukemic patients receiving chemotherapy for at least one cycle and their mean ages 37.1 ± 4.89 years.The patients were selected from National Cancer Institute, Cairo ( inpatient ward). The study lasted from March 2018 to June 2018. Patients were randomly assigned into two groups.Group A (30 patients) who received inspiratory muscles training for 4 successive weeks, 5 sessions/week; and Group B (10 patients) acted as a control group on chemotherapy only. Data obtained from both groups regarding (MVV), 2 min walk test and Quality of life questionnaire (FACT-G) were statistically analyzed and compared

ELIGIBILITY:
Inclusion Criteria:

* male patient with age ranges from 30-50 years
* All patients were leukemic receiving chemotherapy for at least one cycle as a treatment of malignant tumor
* All patients were hemodynamically stable
* All patients were ambulant

Exclusion Criteria:

* lung cancer
* History of any pulmonary disease.
* Metastasis of lungs, ribs, mediastinal structure
* Pulmonary pathology(e.g acute respiratory distress syndrome or exacerbation of chronic obstructive pulmonary disease)
* ruptured ear drum or any other condition of the ear
* High peak airway pressure (barotraumas)
* patients with marked elevated left ventricular end diastolic volume and pressure
* patients with worsening heart failure signs and symptoms

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary ventilation | change from baseline maximum voluntary ventilation at 4 weeks
  It was performed by breathing deeply and rapidly for 10 to 15 seconds using spirometer
2 min walk test | change from baseline 2 min walk test at 4 weeks
  Each patient was asked to cover as much ground as possible over 2 minutes
FACT-G questionnaire | change from baseline FACT-G questionnaire at 4 weeks
  27 questions with four domains assessing physical well being,social well being, emotional well being and functional wellbeing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided